CLINICAL TRIAL: NCT02456155
Title: Study to Compare the Placement Method of Nasal Jejunal Tube in Patients With Severe Acute Pancreatitis: Bedside Placement With Ultrasound Confirmation Versus Placement Endoscopically
Brief Title: A Trial of Bedside Placement of Nasal Jejunal Tube Confirmed by Ultrasound Compared to Placement by Endoscope in Patients With SAP
Acronym: SAP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Gang (Other)
Responsible Party: Sponsor-Investigator, Li Gang, Jinling Hospital, Nanjing University
Organization: Nanjing University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110-92
Record Dates: First submitted 2015-05-05; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Bedside Placement of Nasal Jejunal Tube
Keywords: bedside placement; nasal jejunal tube; ultrasound; severe acute pancreatitis; endoscope; efficacy; safety
MeSH Terms: conditions — Pancreatitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasound group (Experimental): using B ultrasound as a instruction technique to place Nasal Jejunal Tube
  Interventions: Procedure: placing nasal jejunal tube with ultrasound
- endoscope group (Placebo Comparator): Conventional methods for placing Nasal Jejunal Tube
  Interventions: Procedure: placing nasal jejunal tube endoscopically

INTERVENTIONS:
Procedure: placing nasal jejunal tube with ultrasound — bedside placing nasal jejunal tube with ultrasound confirmation versus placing endoscopically
  Arms: ultrasound group
Procedure: placing nasal jejunal tube endoscopically
  Arms: endoscope group

SUMMARY:
The investigators assessed the utility of ultrasonography in confirming the position of nasal jejunal tube after bedside placement when compared with endoscopic placement in patients with severe acute pancreatitis.

Primary endpoint:

Success rate.

Secondary Endpoint:

Adverse effects, Change of intra-abdominal pressure (1h before, 1h after and 3 days after placement), Tolerance of enteral nutrition, Time to approach the target calories.

DETAILED DESCRIPTION:
We set this randomised trial to assess the safety and utility of ultrasonography in confirming the position of nasal jejunal tube after bedside placement when compared with endoscopic placement in patients with severe acute pancreatitis.

Primary endpoint:

Success rate.

Secondary Endpoint:

Adverse effects, Change of intra-abdominal pressure (1h before, 1h after and 3 days after placement), Tolerance of enteral nutrition, Time to approach the target calories.

ELIGIBILITY:
Inclusion Criteria:

* acute pancreatitis patients who need enteral nutrition;
* patients in acute phase of pancreatitis (within 2 weeks from onset);
* the severity of pancreatitis is equal to or above moderate (according to the revised classification of pancreatitis).

Exclusion Criteria:

* diagnosed with IAH(Intra-abdominal pressure) IV grade, abdominal compartment syndrome (ACS);
* patients who have circulatory failure;
* patients who have gastrointestinal bleeding;
* patients who have specific diseases such as chronic digestive diseases and autoimmune diseases;
* patients in pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 24 hours
  Success rate is defined as the right position of nasal jejunal tube confirmed by X-ray.

SECONDARY OUTCOMES:
Adverse effects | 24 hours
  gastrointestinal perforation, gastrointestinal bleeding, tie of the tube, blocking of the tube
Change of intra-abdominal pressure | 3 days
  the intra-abdominal pressure at 1h before, 1h after and 3 days after placement
Tolerance of enteral nutrition | 3 days
  nausea, vomiting, diarrhea, abdominal pain
Time interval to approach the target calories | 7 days
  The exact time interval from the placement of the tube to the time that the patient can tolerate the target enteral nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- JinLing hospital, Nanjing, Jiangsu, China